CLINICAL TRIAL: NCT04731935
Title: A Pilot Study to Evaluate Safety and Efficacy of a Novel Electrode Configuration for Delivering Transcutaneous Auricular Neurostimulation to Improve Symptoms Associated With Opioid Withdrawal
Brief Title: Novel Earpiece for Transcutaneous Auricular Neurostimulation (tAN) for Symptoms of Opioid Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBM-OWP-04
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-01

CONDITIONS: Opioid-use Disorder; Opioid Withdrawal
Keywords: auricular neurostimulation; vagus nerve stimulation; transcutaneous; withdrawal symptoms
MeSH Terms: conditions — Opioid-Related Disorders; Substance Withdrawal Syndrome

STUDY DESIGN:
Intervention Model Description: This study is designed as a pilot, single-center, non-randomized, uncontrolled, clinical trial in which subjects will be consented, receive a baseline assessment and receive tAN treatment and assessment every day during their 3 to 5-day detox treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- tAN Therapy (Experimental): tAN will be delivered at a duty cycle of for 5 minutes ON and 10 seconds OFF for a total of 120 hours (5 days) therapy duration. Stimulation intensity will be customized to the participants comfort level and within range of therapeutic effectiveness.
  Interventions: Device: Sparrow Therapy System

INTERVENTIONS:
Device: Sparrow Therapy System — Transcutaneous auricular neurostimulation

SUMMARY:
The objective of this study is to evaluate whether tAN via the tragus (vagal) and auriculotemporal (trigeminal) nerve pathways results in a clinically meaningful reduction in opioid withdrawal symptoms.

DETAILED DESCRIPTION:
This study is designed as a pilot, single-center, non-randomized, uncontrolled, clinical trial in which subjects will be consented, receive a baseline assessment, and receive tAN treatment and assessment every day during their 3 to 5-day detox treatment. Use of opioid-based medication assisted therapy (MAT) will not be permitted at any point during the study. Use of non-opioid-based MATs (i.e. comfort or rescue medications) will not be permitted until after the subject has completed the 60 minute COWS assessment to ensure changes in COWS score at 60 minutes are only the result of tAN therapy.

ELIGIBILITY:
Inclusion Criteria:

* Current opioid dependence; prescriptive or non-prescriptive
* COWS score is ≥ 13 or in the opinion of the investigator the subject is in moderate to severe withdrawal
* 18-65 years of age
* English proficiency
* Participants must be able to provide informed consent and function at an intellectual level sufficient for study requirements

Exclusion Criteria:

* Current evidence of an uncontrolled and/or clinically significant medical condition
* History of seizures or epilepsy
* History of neurological diseases or traumatic brain injury
* Participants using long-acting opioids such as methadone or buprenorphine for a period of five or more consecutive days prior to enrollment
* Recent suicide attempt leading to current hospital admission or continued expressed suicidal ideation
* Presence of devices (e.g., pacemakers, cochlear prosthesis, neurostimulators)
* Abnormal ear anatomy or ear infection present
* Women of childbearing potential not using adequate contraception as per investigator judgement or not willing to comply with contraception for the duration of the study
* Females who are pregnant or lactating
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Clinical opiate withdrawal scale (COWS) score | 60 minutes
  Mean percent change in clinical opiate withdrawal scale (COWS) score from baseline to 60 minutes after start of tAN therapy. The COWS is an 11-item scale with a score range between 0 and 48. Total score is the sum of all the items and a higher score indicates more severe withdrawal symptoms. Scores between 5 and 12 indicate mild withdrawal, scores between 13 and 24 indicate moderate withdrawal, scores between 25 and 36 indicate moderately severe withdrawal and scores greater than 36 indicate severe withdrawal. A COWS score reduction of 15% or greater for a given individual is considered clinically significant.

SECONDARY OUTCOMES:
Clinical opiate withdrawal scale (COWS) score | 30 minutes
  Mean percent change in COWS score from baseline to 30 minutes after start of tAN therapy.
Clinical opiate withdrawal scale (COWS) score | 120 minutes
  Mean percent change in COWS score from baseline to 120 minutes after start of tAN therapy.
Clinical opiate withdrawal scale (COWS) score | Days 2-5
  Mean percent change in COWS score from baseline to Days 2 through 5 after start of tAN therapy.

OTHER OUTCOMES:
Heart rate variability measured by R to R interval | Days 2-5
  Mean change from baseline to Days 2-5 in heart rate variability measured by R to R interval.
Patient Health Questionnaire (PHQ-9) | Day 5
  Mean change in depression symptoms measured by Patient Health Questionnaire (PHQ-9) total score from baseline to Day 5. The PHQ-9 is a nine-item depression scale based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. Each of the nine items is rated on a 0 (not at all) to 3 (nearly every day) scale. A total score is calculated by summing the nine items. Scores range from 0 to 27 and higher scores indicate a higher degree of depression.
Post-Traumatic Stress Disorder (PTSD) Checklist for DSM-5 (PCL-5) | Day 5
  Mean change in PTSD symptoms measured by the PTSD Checklist for DSM-5 (PCL-5) total symptom severity score from baseline to Day 5. The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Each of the 20 items is rated on a 0 (not at all) to 4 (extremely) scale. A total symptom severity score is calculated by summing the 20 items. Scores range from 0 and 80 and higher scores indicating a higher degree of PTSD symptomology. Evidence suggests that a10-20 point reduction in score represents a clinically significant change in PTSD symptoms.
World Health Organization Quality of Life - BREF (WHOQOL-BREF) | Day 5
  Mean change in WHOQOL-BREF domain scores (physical health, psychological health, social relationships, environment, and overall QoL/general health) from baseline to Day 5. The World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a 26-item, self-report questionnaire which assesses 4 quality of life domains: physical health, psychological health, social relationships, and environment. In addition, there are 2 items that measure overall quality of life and general health. Subjects rate how much they have experienced each item in the preceding 2 weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely). Domain scores are scaled in a positive direction with higher scores denoting higher quality of life. Raw domain scores will be converted to a 0 to 100 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Navid Khodaparast, PhD, Study Director — Spark Biomedical, Inc.
Locations (1):
- Recovery Unplugged, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No